CLINICAL TRIAL: NCT06419998
Title: One Stage Transanal Versus One Stage Laparoscopic-assisted Transanal Endorectal Pull-through in the Management of Hirschsprung's Disease in Pediatric Age Group; A Retrospective Study.
Brief Title: Transanal Versus Laparoscopic-assisted Transanal Through in the Management of Hirschsprung's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Ahmed Elrouby, Associate Professor of pediatric Surgery, Egyptian Biomedical Research Network
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0306356
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Disorder; Hirschprung's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Pediatric patients presented with Hirschsprung's disease treated by pure transanal endorectal pull-through (TAERPT)
  Interventions: Procedure: Group A: Pure transanal endorectal pull-through (TAERPT)
- Group B (Active Comparator): Pediatric patients presented with Hirschsprung's disease treated by laparoscopic-assistance endorectal pull-through (LAERPT)
  Interventions: Procedure: Group B: Laparoscopic-assistance endorectal pull-through (LAERPT)

INTERVENTIONS:
Procedure: Group A: Pure transanal endorectal pull-through (TAERPT) — Patients of Group A will be treated totally by pure transanal endorectal pull-through without the assistance of laparoscopy
  Arms: Group A
Procedure: Group B: Laparoscopic-assistance endorectal pull-through (LAERPT) — Patients of Group B will be treated transanal endorectal pull-through but with the assistance of laparoscopy
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare the surgical and functional outcomes of pure transanal endorectal pull-through (TAERPT) and laparoscopic-assistance endorectal pull-through (LAERPT) in pediatric patients presented with Hirschsprung's Disease between 3 months and 18 years old.

The main questions our study aims to answer are:

* Does post-operative continence differs between the two groups?
* Does post-operative constipation differs between the two groups?
* Does post-operative soiling differs between the two groups
* Does post-operative enterocolitis differs between the two groups?
* Do post-operative complications differ between the two groups? If there is a comparison group: Researchers will compare between pure transanal endorectal pull-through (TAERPT) and laparoscopic-assistance endorectal pull-through (LAERPT) to see if there is a difference in post-operative continence, constipation, soiling, enterocolitis or complications.

Participants will be divided into two groups; 40 patients will be treated by TAERPT and included in Group A and 30 patients will be treated by LAERPT and included in Group B.

DETAILED DESCRIPTION:
Introduction: One-stage treatment of endorectal pull-through for Hirschsprung's disease could be approached through a complete transanal approach or with the assistance of laparoscopy. Our study aims to compare the surgical and functional outcomes of pure transanal endorectal pull-through (TAERPT) and laparoscopic-assistance endorectal pull-through (LAERPT). Material & methods: This retrospective study included 70 pediatric patients presented with Hirschsprung's Disease to Elshatby University Hospital. 40 patients were treated by TAERPT and included in Group A and 30 patients were treated by LAERPT and included in Group B. The two groups were compared as regards the operative data as well as the post-operative outcomes including the time of passage of stools, time of tolerating oral feeding, the duration of hospital stay, and the development of any early postoperative complications. Also, the number of bowel habits, constipation, enterocolitis, abdominal distension, anastomotic stricture, and continence were assessed.

ELIGIBILITY:
Inclusion Criteria

* Pediatric patients with age range between 3 months and 18 years old presented with Hirschsprung's Disease who were confirmed to have this condition by contrast enema and/or rectal biopsy.

Exclusion Criteria:

* Patients with previous colostomy.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Post-operative continence | One post-operative year
  The two groups will be compared according to post-operative continence whether continent or incontinent by using Abbreviated Baylor Social Continence Scale. the sore ranges from 0 to 24 with the minimum score revealing an excellent result and the highest score revealing the worst result. (Excellent = 0-5, Good = 7-12, Fair = 13-18, Poor = 19-24)
Post-operative constipation | One post-operative year
  The two groups will be compared according to post-operative constipation whether present or not
Post-operative soiling | One post-operative year
  The two groups will be compared according to post-operative soiling whether present or not
Post-operative enterocolitis | One post-operative year
  The two groups will be compared according to post-operative enterocolitis whether present or not
Post-operative complications | One post-operative year
  The two groups will be compared according to post-operative complications whether present or not

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed El Rouby, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elrouby A, Shehata S, Waheeb S, Khairi A, AbdAl-Aziz D, Looka B. One stage transanal versus one stage laparoscopic-assisted transanal endorectal pull-through in managing Hirschsprung's disease in pediatric age group; a retrospective study. BMC Surg. 2025 Feb 8;25(1):59. doi: 10.1186/s12893-025-02768-1. PMID 39922991